CLINICAL TRIAL: NCT03731572
Title: Hip Muscle Power, Lateral Balance Function, and Falls in Aging
Acronym: HIPS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: VA Maryland Health Care System (U.S. Federal Agency)
Responsible Party: Principal Investigator, Vicki Gray, Assistant Professor, University of Maryland, Baltimore
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Prevention
Other Study IDs: HP-00082488
Record Dates: First submitted 2018-10-01; First posted 2018-11-06 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Accidental Falls
Keywords: Falls; Balance; Protective Stepping; Lateral Balance; Elderly; Power training
MeSH Terms: interventions — Resistance Training

STUDY DESIGN:
Intervention Model Description: The investigators will compare changes in protective stepping, hip abduction and adduction muscle power and neuromuscular activation, balance and mobility function, and number of prospective falls between power and strength training groups.
Who Masked: Investigator, Outcomes Assessor
Masking Description: All testing for Aims 1a and 1b will be conducted by individuals who are masked to subject intervention group assignment at baseline-testing, post-intervention testing, and retention-testing
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Power Training (Experimental): Hip abductor-adductor resistance exercises at 75% maximum strength and maximum execution speed, 3, 1-hour training sessions per week for 12 weeks.
  Interventions: Other: Power Training
- Strength Training (Active Comparator): Hip muscle abductor-adductor resistance exercises at maximum strength at reduced execution speed (2s concentric/3s eccentric), 3, 1-hour training sessions per week for 12 weeks.
  Interventions: Other: Strength Training

INTERVENTIONS:
Other: Power Training — Hip abductor-adductor resistance exercises at maximum execution speed
  Arms: Power Training
Other: Strength Training — Hip abductor-adductor resistance exercises at reduced execution speed
  Arms: Strength Training

SUMMARY:
Falls and their consequences are among the major problems in the medical care of older individuals. The long-term goal of this research is to develop a mechanistically based therapeutic intervention to enhance muscle power, weight-shifting capability, and lateral balance function through protective stepping to prevent falls. When human balance is challenged, protective stepping is a vital strategy for preventing a fall during activities of daily life. Many older people at risk for falls have particular difficulties with successfully stepping sideways as a protective response to loss of balance in the lateral direction. Age-related declines in lateral balance function result from neuromuscular and biomechanical limitations in hip abductor-adductor muscle power generation. This study will test whether these impairments can be improved with high-velocity hip muscle resistance power training that will be more effective than conventional resistance strength training.

DETAILED DESCRIPTION:
Falls and their consequences are among the major problems in the medical care of older individuals. The long-term goal of this research is to develop a mechanistically based therapeutic intervention to enhance muscle power, weight-shifting capability, and lateral balance function through protective stepping to prevent falls. When human balance is challenged, protective stepping is a vital strategy for preventing a fall during activities of daily life. Many older people at risk for falls have particular difficulties with successfully stepping sideways as a protective response to loss of balance in the lateral direction. The investigators propose that age-related declines in lateral balance function through impaired weight transfer and protective stepping linked with falls, result from neuromuscular and biomechanical limitations in hip abductor-adductor (AB-AD) muscle power generation. Moreover, the investigators hypothesize that these balance and neuromotor impairments can be improved with high-velocity muscle resistance power training that will be more effective than conventional muscle resistance strength training. The specific aims are, Aim 1: To conduct a single blind, randomized, and controlled trial comparing the effects of 12 weeks of hip AB-AD muscle power training against strength training, and the rate of retention after 3 months of no training in community living older adults by determining a) the changes in neuromotor performance (kinetics, kinematics, muscle activation patterns) of pre-step weight transfer during waist-pull induced side stepping, and rapid voluntary reaction time (RT) sidestepping; and by b) the changes in isolated hip AB-AD muscle neuromotor performance. Weight shifting and stepping ability will be tested with different initial induced stepping limb load conditions, and by varying voluntary stepping limb selection certainty with simple and choice RT tasks; Aim 2: To compare the effectiveness of hip AB-AD muscle power and strength training in reducing the rate of prospective falls over a one-year monitoring period post-training. Secondary analyses will assess the number of in-task falls, and the effect of muscle power versus strength training on changes in functional balance and mobility. Overall, the studies are expected to establish support for the superiority of velocity dependent power training over strength training on enhancing muscle performance, protective balance control and functional mobility outcomes, and for the prevention of falls among older adults.

ELIGIBILITY:
Inclusion Criteria:

1. 65 years of age or older
2. Functionally independent
3. Living in the community
4. Generally healthy

Exclusion Criteria:

1. Cognitive impairment (Mini Mental Score Exam less than 24)
2. Sedative use
3. Non-ambulatory
4. Any clinically significant musculoskeletal impairment
5. Any clinically significant neurological impairment
6. Any clinically significant cardiopulmonary impairment
7. Any clinically significant metabolic impairment
8. Any general medical problem that will interfere with testing or training
9. Diabetes, renal, or liver disease by identified by routine chemistry

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 97 (Actual)
Dates: Start 2019-09-16 (Actual); Primary Completion 2026-01-10 (Actual); Study Completion 2026-01-10 (Actual)

PRIMARY OUTCOMES:
Incidence of single lateral steps | At 3 months
  Change in number of single steps between pre and post tests

SECONDARY OUTCOMES:
Hip muscle power | At 3 months
  Change in maximum hip power between pre and post tests
Number of Falls | 12 months
  Total number of falls reported at 1 year follow up.

CONTACTS AND LOCATIONS:
Overall Officials: Vicki L Gray, PhD, Principal Investigator — University of Maryland, Baltimore
Locations (1):
- VA Maryland Health Care System, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No